CLINICAL TRIAL: NCT01056588
Title: Predictors of Smoking Outcomes During Treatment Programs
Brief Title: Contingency Management for Smoking Abstinence With Adolescent Smokers
Acronym: CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: University of Florida (Other)
Responsible Party: Principal Investigator, Brady Reynolds, Associate Professor, University of Kentucky
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB09-00399
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Cigarette Smoking
Keywords: adolescent smoking; Contingency management; Quit smoking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Condition (Placebo Comparator): In this condition, participants will receive reinforcement for timely breath samples with no contingency for a specific breath CO level.
  Interventions: Behavioral: Control condition
- CO-Contingent (Active Comparator): In this condition, participants will receive reinforcements contingent on submitting breath samples at CO levels indicating reductions or abstinence from smoking.
  Interventions: Behavioral: CO-Contingent

INTERVENTIONS:
Behavioral: CO-Contingent — In this 42 day condition, participants will receive monetary reinforcements contingent on submitting breath samples at CO levels indicating reductions or abstinence from smoking (4ppm).
  Arms: CO-Contingent
Behavioral: Control condition — In this condition, participants will receive monetary reinforcement for timely breath samples with no contingency for a specific breath CO level
  Arms: Control Condition

SUMMARY:
The primary objective of this research is to evaluate the effectiveness of this type of smoking cessation program by comparing a treatment group with a control group.

A secondary objective of this research is to explore relations between impulsive behavior and smoking-cessation success among treatment-seeking teens participating in a quit-smoking program.

Hypothesis 1. A greater proportion of the participants in the treatment condition will be verified as abstinent from smoking during the course of treatment than participants of the control condition.

Hypothesis 2. It is hypothesized that teens who do not successfully stop smoking (or who drop out of the treatment program) will be more impulsive (from measures taken just prior to treatment) than those who do successfully stop or significantly reduce rate of smoking.

DETAILED DESCRIPTION:
In response to the need for treatments appropriate for adolescent smokers, this research (utilizing a two-group randomized-control design, n = 63 per group) will evaluate the effectiveness and efficacy of a new and innovative Internet-based contingency-management (CM) program for smoking abstinence with adolescent smokers. This program lasts for 42 days and involves a 21 day abstinence phase. For the treatment condition, participants are reinforced for breath samples that verify abstinence from smoking three times per day; however, for the control condition, participants are reinforced for timely breath samples regardless of abstinence status.

Because this CM program is Internet based it can be completed from home, which stands to be more viable as a treatment option for adolescent smokers than other treatments requiring frequent trips to a clinical facility. From preliminary work with adult and adolescent smokers, it is expected this treatment program will be highly effective in creating favorable changes in adolescent smoking behavior. This research will also involve eight monthly post-treatment follow-up sessions to determine long-term consistencies or changes in smoking behavior.

A secondary goal of this research is to explore pre-treatment assessments of different dimensions of impulsive behavior as predictors of treatment outcome. These behavioral assessments will provide highly detailed information about the specific behavioral styles of adolescent smokers who are unable to effectively change their smoking behavior during treatment. This information should provide new points of emphasis for treatment-program modifications to improve these programs to be more effective for adolescents most challenged in their efforts to quit or reduce smoking.

ELIGIBILITY:
Inclusion Criteria:

* Ages of 13-19
* Have a breath CO level of at least 10ppm
* Smoke at least 2 cigarettes per day
* Live in Columbus, OH area

Exclusion Criteria:

* Adolescents must be English-speaking

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 126 (Actual)
Dates: Start 2010-02 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome for this research will be smoking treatment outcomes (reductions or abstinence) compared across the treatment- and control-condition arms. | approximately 9.5 months

SECONDARY OUTCOMES:
The secondary outcome for this research will involve the use of pre-treatment assessments of impulsive behavior as predictors of treatment response at the end of the treatment for both conditions and also during followup. | approximately 9.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Brady Reynolds, PhD, Principal Investigator — Nationwide Children's Hopsital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States